CLINICAL TRIAL: NCT00569582
Title: An Open-label Study of the Efficacy and Safety of CORLUX (Mifepristone) in the Treatment of the Signs and Symptoms of Endogenous Cushing's Syndrome
Brief Title: A Study of the Efficacy and Safety of CORLUX in the Treatment of Endogenous Cushing's Syndrome
Acronym: SEISMIC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-1073-400
Record Dates: First submitted 2007-12-05; First posted 2007-12-07 (Estimated); Results first posted 2012-05-28 (Estimated); Last update posted 2013-08-22 (Estimated); Status verified 2013-08

CONDITIONS: Cushing's Syndrome
Keywords: Cushing's Disease; Cushing's Syndrome; Cushings; Pituitary; ACTH; Adrenocorticotropic hormone; Ectopic; Adrenal adenoma; Adrenal carcinoma; Adrenal autonomy; Cortisol; Hypercortisolemia; Cushingoid; Moon facies; Dorsocervical fat; Plethora; Hirsutism; Violaceous striae; Hormone; Contraceptive; Endocrine; Cushing Syndrome; Ectopic ACTH Secretion
MeSH Terms: conditions — Cushing Syndrome; Pituitary ACTH Hypersecretion; Pituitary Diseases; Choristoma; ACTH Syndrome, Ectopic; Adrenal Cortex Neoplasms; Hirsutism | interventions — Mifepristone; Corlux

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: mifepristone

INTERVENTIONS:
Drug: mifepristone — Patients take mifepristone by mouth once a day. The dose is increased during scheduled timepoints during the study or until symptoms improve or the highest dosage allowed is reached. Dose escalation will be based upon weight. During clinic visits, blood pressure, glucose tolerance and blood chemistries are measured and EKG and urinalysis will be performed.
  Other Names: CORLUX

SUMMARY:
Patients will receive Corlux (mifepristone) daily for up to 24 weeks. Assessments of the signs and symptoms of Cushing's syndrome will be obtained.

DETAILED DESCRIPTION:
Cushing's syndrome is a relatively rare disorder caused by prolonged exposure to high levels of the glucocorticoid hormone cortisol. Cushing's syndrome may result from elevated endogenous or exogenous sources of cortisol. Endogenous Cushing's syndrome resulting from cortisol overproduction by the adrenal glands is the subject of this protocol. Patients with exogenous Cushing's syndrome, which develops as a side effect of chronic administration of high doses of glucocorticoids, are not eligible for enrollment in this study.

This will evaluate the safety and efficacy of mifepristone for treatment of the signs and symptoms of hypercortisolemia in patients with endogenous Cushing's syndrome from ACTH-dependent or adrenal disorders.

The study will enroll subjects for whom the investigator has determined that medical treatment of endogenous hypercortisolemia is needed. Medical treatment may be intended to treat the effects of persistent or recurrent hypercortisolemia after surgery and/or radiation for Cushing's syndrome, to bridge the period of time for radiation to become effective, or when surgery is not feasible.

ELIGIBILITY:
Inclusion Criteria:

Individuals eligible for enrollment into this study are adult male and non-pregnant female adult patients who:

* Are at least 18 years of age
* Have a confirmed diagnosis of endogenous hypercortisolemia caused by ACTH dependent or ACTH independent etiologies, including

  1. Cushing's Disease (that has recurred after primary pituitary surgery, or has failed pituitary surgery, or has been treated with radiation therapy to the pituitary, or is not treatable with surgery, or exists in patients who are not candidates for surgery, and is confirmed by documentation of ACTH immuno-reactivity on a pathological evaluation of pituitary tissue from a previous surgical specimen or IPSS with a central-to-peripheral gradient (ratio) of >2 before or >3 after CRH administration).
  2. Ectopic ACTH
  3. Ectopic CRF secretion
  4. Adrenal adenoma
  5. Adrenal carcinoma
  6. Adrenal autonomy
* Require medical treatment of hypercortisolemia
* Have diabetes mellitus type 2 or glucose intolerance AND/OR have hypertension *Note: To be eligible for inclusion subjects must have documented evidence of persistent endogenous hypercortisolemia

Exclusion Criteria:

Individuals not eligible to be enrolled into the study are those who:

* Have de novo Cushing's disease and are surgical candidates for pituitary surgery.
* Have an acute or unstable medical problem, which could be aggravated by mifepristone treatment.
* Taking medications within 14 days of the baseline visit (Day 1) that a) have a large first pass metabolism largely mediated by CYP3A4 and a narrow therapeutic margin and/or b) are strong CYP3A4 inhibitors.
* Female patients of reproductive potential, who are pregnant or who are unable or unwilling to use medically acceptable, non-hormonal methods of contraception during the study.
* Have received investigational treatment (drug, biological agent or device) within 30 days of Screening
* Have a history of an allergic reaction or intolerance to CORLUX (mifepristone)
* Have a non-endogenous source of hypercortisolemia such as factious hypercortisolemia (exogenous source of glucocorticoid, iatrogenic Cushing's syndrome), factious or therapeutic use of ACTH
* Have Pseudo-Cushing's syndrome.
* Receive PPARgamma agonist drugs (e.g. pioglitazone, rosiglitazone) within 4 months of Baseline (Day 1).
* Postmenopausal women with an intact uterus who have experienced unexplained vaginal bleeding within 12 months of Screening are excluded.
* Have renal failure as defined by a serum creatinine of ≥2.2 mg/dL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-12; Primary Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Coleman Gross, Study Director — Corcept Therapeutics
Locations (17):
- United States (17):
  - University of Alabama at Birmingham School of Medicine, Birmingham, Alabama
  - AMCR Institute Inc., Escondido, California
  - Stanford University Medical Center, Stanford, California
  - The Center for Diabetes and Endocrine Care, Hollywood, Florida
  - Northwestern University Feinberg Medical; Division of Endocrinology, Metabolism & Molecular Medicine, Chicago, Illinois
  - The University of Chicago, Chicago, Illinois
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of New Mexico HSC, Albuquerque, New Mexico
  - Cleveland Clinic Foundation; Dept of Endocrinology, Diabetes & Metabolism, Cleveland, Ohio
  - Oklahoma University Health Science Center, Oklahoma City, Oklahoma
  - Oregon Health Sciences University, Portland, Oregon
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Diabetes and Glandular Disease Clinic, San Antonio, Texas
  - Endocrinology Center at North Hills, Froedtert and Medical College of Wisconsin, Menomonee Falls, Wisconsin

REFERENCES:
- [Background] Sartor O, Cutler GB Jr. Mifepristone: treatment of Cushing's syndrome. Clin Obstet Gynecol. 1996 Jun;39(2):506-10. doi: 10.1097/00003081-199606000-00024. PMID 8734015
- [Background] Johanssen S, Allolio B. Mifepristone (RU 486) in Cushing's syndrome. Eur J Endocrinol. 2007 Nov;157(5):561-9. doi: 10.1530/EJE-07-0458. PMID 17984235
- [Background] Morris D, Grossman A. The medical management of Cushing's syndrome. Ann N Y Acad Sci. 2002 Sep;970:119-33. doi: 10.1111/j.1749-6632.2002.tb04418.x. PMID 12381547
- [Background] Chu JW, Matthias DF, Belanoff J, Schatzberg A, Hoffman AR, Feldman D. Successful long-term treatment of refractory Cushing's disease with high-dose mifepristone (RU 486). J Clin Endocrinol Metab. 2001 Aug;86(8):3568-73. doi: 10.1210/jcem.86.8.7740. PMID 11502780
- [Background] Agarwai MK. The antiglucocorticoid action of mifepristone. Pharmacol Ther. 1996;70(3):183-213. doi: 10.1016/0163-7258(96)00016-2. PMID 8888066
- [Background] Miller JW, Crapo L. The medical treatment of Cushing's syndrome. Endocr Rev. 1993 Aug;14(4):443-58. doi: 10.1210/edrv-14-4-443. No abstract available. PMID 7693447
- [Background] Nieman LK, Chrousos GP, Kellner C, Spitz IM, Nisula BC, Cutler GB, Merriam GR, Bardin CW, Loriaux DL. Successful treatment of Cushing's syndrome with the glucocorticoid antagonist RU 486. J Clin Endocrinol Metab. 1985 Sep;61(3):536-40. doi: 10.1210/jcem-61-3-536. PMID 2991327
- [Result] Fleseriu M, Biller BM, Findling JW, Molitch ME, Schteingart DE, Gross C; SEISMIC Study Investigators. Mifepristone, a glucocorticoid receptor antagonist, produces clinical and metabolic benefits in patients with Cushing's syndrome. J Clin Endocrinol Metab. 2012 Jun;97(6):2039-49. doi: 10.1210/jc.2011-3350. Epub 2012 Mar 30. PMID 22466348
- [Derived] Fein HG, Vaughan TB 3rd, Kushner H, Cram D, Nguyen D. Sustained weight loss in patients treated with mifepristone for Cushing's syndrome: a follow-up analysis of the SEISMIC study and long-term extension. BMC Endocr Disord. 2015 Oct 27;15:63. doi: 10.1186/s12902-015-0059-5. PMID 26507877
- [Derived] Fleseriu M, Findling JW, Koch CA, Schlaffer SM, Buchfelder M, Gross C. Changes in plasma ACTH levels and corticotroph tumor size in patients with Cushing's disease during long-term treatment with the glucocorticoid receptor antagonist mifepristone. J Clin Endocrinol Metab. 2014 Oct;99(10):3718-27. doi: 10.1210/jc.2014-1843. Epub 2014 Jul 11. PMID 25013998
- [Derived] Wallia A, Colleran K, Purnell JQ, Gross C, Molitch ME. Improvement in insulin sensitivity during mifepristone treatment of Cushing syndrome: early and late effects. Diabetes Care. 2013 Sep;36(9):e147-8. doi: 10.2337/dc13-0246. No abstract available. PMID 23970725
- See also: Corporate Website — http://www.corcept.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 24 week multicenter, open-label trial after failed multimodality therapy at 14 U.S. academic medical centers and three private research centers.
Pre-assignment Details: Adults with endogenous Cushing's Syndrome associated with either type 2 diabetes mellitus/impaired glucose tolerance or a diagnosis of hypertension.
Groups:
- Mifepristone: Mifepristone was administered at doses of 300-1200 mg daily.
Period: Overall Study
Arm/Group | Mifepristone
Started | 50
Completed | 34
Not Completed | 16
Not completed — Withdrawal by Subject | 5
Not completed — Death | 2
Not completed — Adverse Event | 7
Not completed — Subject was too ill to travel. | 1
Not completed — Subject was non-compliant. | 1

BASELINE CHARACTERISTICS:
Arm/Group | Mifepristone
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 46
  >=65 years | 4
Age Continuous [Mean (Standard Deviation); unit: years] | 45.4 (11.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Diabetes and/or Glucose Intolerance.
Description: Responder is defined as subject with a decrease greater than or equal to 25% in area under the curve for glucose on 2-hour oral glucose test from baseline to week 24 or last visit, for Cushing's patients with type-2 diabetes mellitus/impaired glucose tolerance.
Time Frame: Baseline to Week 24
Population: Patients with at least 30 days of dosing.
Measure: Number; unit: participants
Arm/Group | Mifepristone
Number analyzed (Participants) | 25
participants | 15

2. Primary Outcome: Decrease in Diastolic Blood Pressure.
Description: Responder is defined as subject with a decrease greater than or equal to 5mm Hg in diastolic blood pressure from baseline to week 24 or last visit.
Time Frame: Baseline to Week 24
Measure: Number; unit: participants
Arm/Group | Mifepristone
Number analyzed (Participants) | 21
participants | 8

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Mifepristone
Serious Adverse Events (participants affected / at risk) | 16/50
Other Adverse Events (participants affected / at risk) | 49/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mifepristone (N=50)
Legionella pneumonia (Infections and infestations) | 1 (1)
Gastritis Erosive (Gastrointestinal disorders) | 1 (1)
Foot Fracture (Injury, poisoning and procedural complications) | 1 (1)
Intracranial Aneurysm (Nervous system disorders) | 1 (1)
Orthostatic Hypotension (Vascular disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Confusional State (Psychiatric disorders) | 1 (1)
Blood Potassium Decreased (Investigations) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 1 (1)
Renal Failure Acute (Renal and urinary disorders) | 1 (1)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) — severe
Sinusitis (Infections and infestations) | 1 (1)
Asthenia (General disorders) | 1 (2)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Adrenal Insufficiency (Endocrine disorders) | 1 (1)
Subcutaneous Abscess (Infections and infestations) | 1 (1)
Angina Pectoris (Cardiac disorders) | 1 (1)
adrenal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Mifepristone (N=50)
Nausea (Gastrointestinal disorders) | 24 (40)
Vomiting (Gastrointestinal disorders) | 13 (21)
Dry mouth (Gastrointestinal disorders) | 9 (12)
Diarrhoea (Gastrointestinal disorders) | 6 (8)
Constipation (Gastrointestinal disorders) | 5 (5)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 (4)
Fatigue (General disorders) | 24 (37)
Oedema peripheral (General disorders) | 13 (31)
Pain (General disorders) | 7 (9)
Asthenia (General disorders) | 3 (5) — mild
Malaise (General disorders) | 3 (4)
Oedema (General disorders) | 3 (6)
Pitting oedema (General disorders) | 3 (4)
Thirst (General disorders) | 3 (3)
Headache (Nervous system disorders) | 22 (40)
Dizziness (Nervous system disorders) | 11 (20)
Somnolence (Nervous system disorders) | 5 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 (20)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (9)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (11)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (6)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 (6)
Flank pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Blood potassium decreased (Investigations) | 17 (27)
Thyroid function test abnormal (Investigations) | 9/18 (11)
Blood triglycerides increased (Investigations) | 4 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (5)
Ecchymosis (Skin and subcutaneous tissue disorders) | 4 (4)
Acne (Skin and subcutaneous tissue disorders) | 3 (5)
Sinusitis (Infections and infestations) | 7 (9)
Nasopharyngitis (Infections and infestations) | 6 (10)
Urinary tract infection (Infections and infestations) | 4 (5)
Upper respiratory tract infection (Infections and infestations) | 3 (5)
Decreased appetite (Metabolism and nutrition disorders) | 10/20 (12)
Anorexia (Metabolism and nutrition disorders) | 5 (6)
Hypoglycaemia (Metabolism and nutrition disorders) | 3 (4)
Hypertension (Metabolism and nutrition disorders) | 12 (14)
Hot flush (Metabolism and nutrition disorders) | 3 (3)
Vaginal haemorrhage (Reproductive system and breast disorders) | 4 (4)
Metrorrhagia (Reproductive system and breast disorders) | 3 (8)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (11) — mild or moderate
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Anxiety (Psychiatric disorders) | 5 (12)
Insomnia (Psychiatric disorders) | 3 (5)
Contusion (Injury, poisoning and procedural complications) | 3 (4)
Vision blurred (Eye disorders) | 4 (5)
Cushing's syndrome (Endocrine disorders) | 4 (6)
Pollakiuria (Renal and urinary disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days